CLINICAL TRIAL: NCT04432636
Title: Gut Bacteria and Brain of the Baby: to Link up the Dynamic of Gut Colonization in Preterms Born at Gestational Age of 30-326/7 Weeks and Their Psychomotor Development at 2 Years
Brief Title: Gut Bacteria and Brain of the Baby
Acronym: BaBBa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC19_9784_BaBBa
Record Dates: First submitted 2020-02-19; First posted 2020-06-16 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Premature
MeSH Terms: conditions — Premature Birth | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective French population based cohort (Other): * Data collection of environmental factors at the recruitment
  * Collection of maternal feces
  * Collection of infant feces:
  * A food questionnaire completed by the mother the week after delivery, a food questionnaire on the infant alimentation and food behavior during the period of 2 and 10 months of age, completed by the parents and given to the pediatrician at the medical check-up at the corrected age of 1 year and a food questionnaire on the infant alimentation and food behavior during the period of 12 and 24 months of age, completed by the parents and given to the pediatrician at the medical check-up at the corrected age of 2 years
  * A sample of 15 mL of milk drunk by the preterm at the 7th postnatal day
  * The 'Ages and Stages Questionnaire' ASQ survey completed by the parents and given to the pediatrician at the corrected age of 2 years medical check-up
  Interventions: Other: Data collection of environmental factors; Other: Collection of maternal feces; Other: Collection of infant feces; Other: food questionnaire; Other: a food questionnaire on the infant alimentation and food behavior during the period of 2 and 10 months of age; Other: a food questionnaire on the infant alimentation and food behavior during the period of 12 and 24 months of age; Other: Sample of milk; Other: The 'Ages and Stages Questionnaire' ASQ

INTERVENTIONS:
Other: Data collection of environmental factors — - Data collection of environmental factors (including maternal nutrition and social level, mode of delivery, birth weight, mode of infant feeding, antibiotic treatments) at the recruitment
Other: Collection of maternal feces — - Collection of maternal feces: the first sample after delivery and once a week during the period of hospitalization of their infant (i.e. 5 to 8 samples per mother)
Other: Collection of infant feces — - Collection of infant feces: the first sample after birth and once a week during the period of hospitalization of the baby (i.e. 5 to 8 samples per mother) and a sample collected at the corrected age of 1 year and 2 years (i.e. 8 to 10 samples per infant)
Other: food questionnaire — - A food questionnaire completed by the mother the week after delivery,
Other: a food questionnaire on the infant alimentation and food behavior during the period of 2 and 10 months of age — a food questionnaire on the infant alimentation and food behavior during the period of 2 and 10 months of age, completed by the parents and given to the pediatrician at the medical check-up at the corrected age of 1 year
Other: a food questionnaire on the infant alimentation and food behavior during the period of 12 and 24 months of age — a food questionnaire on the infant alimentation and food behavior during the period of 12 and 24 months of age, completed by the parents and given to the pediatrician at the medical check-up at the corrected age of 2 years
Other: Sample of milk — A sample of 15 mL of milk drunk by the preterm at the 7th postnatal day (if not possible between the 7th and the 10th postnatal days).
Other: The 'Ages and Stages Questionnaire' ASQ — - The 'Ages and Stages Questionnaire' ASQ survey completed by the parents and given to the pediatrician at the corrected age of 2 years medical check-up

SUMMARY:
The project is a prospective French population based cohort. A hundred moderate preterms born at GA30-326/7 will be enrolled for a longitudinal follow-up up to 2 years of corrected age. Eligible neonates will be those born at 30-326/7 weeks of gestation admitted to the neonatal intensive care unit of Rennes Hospital, including transferred infants during the first day of life. The infants will be followed up to the corrected age of 2 years by pediatricians.

ELIGIBILITY:
Inclusion Criteria:

* Preterms born at gestational age of 30-326/7 weeks of amenorrhea
* Preterms born in Rennes hospital or preterms born in another hospital but moved to Rennes hospital during the first 24 h of postnatal life
* Parents or holder of the parental authority who give in writing their free, prior and informed consent for recruitment of their baby who has a social security system
* Mother of the baby who gives in writing her free, prior and informed consent to be involved in the present study
* Mother of the baby who has a social security system

Exclusion Criteria:

* Preterms born with a genetic disease
* Preterms born with a digestive defect
* Uncompetent parents under the protection of guardianship or tutelage services

Ages: 30 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
to associate preterms microbial profiles and psychomotor outcomes at 2 years of corrected age using the 'Ages and Stages Questionnaire' ASQ survey | at 2 years of corrected age
  To associate preterms microbial profiles (bacteria and fungi; alpha- and beta-diversity, abundancies and complex interactions between neonatal microbiotas) and psychomotor outcomes at 2 years of corrected age using the 'Ages and Stages Questionnaire' survey. Each questionnaire includes 30 items covering five developmental domains: communication abilities, gross motor skills, fine motor skills, problem solving abilities, and personal-social skills. Items are scored on a three point scale depending on whether the child performs the task: yes (10 points), sometimes (5 points), or not yet (0 points). Responses are summed to give a score of 0 to 60 for each domain and an overall maximum ASQ score of 300 points. Analyses were based on domain specific scores, using established screening cut-off points: an ASQ score below threshold was defined as a score lower than 2 standard deviations from the mean on any of the five domains.

SECONDARY OUTCOMES:
interactions between maternal and neonatal microbiotas - 2 | at 2 years of corrected age
  Pearson correlation values between maternal microbiota composition and infant gut microbiota composition from birth up to 2 years at corrected age..
interactions between maternal and neonatal microbiotas - 1 | at 1 year of corrected age
  .Pearson correlation values between maternal microbiota composition and infant gut microbiota composition from birth up to 1 year at corrected age.
Bacterial and fongal microbiotas | at 1 year of corrected age
  Pearson correlation values between bacterial (16S) and fongal (18S) microbiota composition in infant from birth up to 1 year at corrected age.
Bacterial and fongal microbiotas | at 2 years of corrected age
  Pearson correlation values between bacterial (16S) and fongal (18S) microbiota composition in infant from birth up to 2 years at corrected age.
maternal dietary profiles and maternal microbiota | up to 8 weeks after delivery
  - Correlation between maternal dietary profiles (food questionnaire completed by the mother the week after delivery) and maternal microbiota. Associations between clinical metadata, dietary profiles and microbial community abundance will be investigate by Multivariate Association with Linear Models (MaAslin).
maternal dietary profiles and maternal microbiota | up to one week after delivery
  - Correlation between maternal dietary profiles (food questionnaire completed by the mother the week after delivery) and maternal microbiota. Associations between clinical metadata, dietary profiles and microbial community abundance will be investigate by Multivariate Association with Linear Models (MaAslin).
maternal dietary profiles and maternal milk composition | at the 7th postnatal day
  - Correlation between maternal dietary profiles (food questionnaire completed by the mother the week after delivery) and maternal milk (a sample of milk drunk by the preterm at the 7th postnatal day, if not possible between the 7th and the 10th postnatal days) composition. The interactions will be assessed by Pearson correlation analysis and drewing the interaction network using Cystoscape package in R.
maternal dietary profiles, maternal milk composition and preterms gut microbiotas | Up to the 2 years of the baby
  - Correlation between maternal maternal dietary profiles (food questionnaire completed by the mother the week after delivery) and maternal milk (a sample of milk drunk by the preterm at the 7th postnatal day, if not possible between the 7th and the 10th postnatal days) composition and preterms gut microbiotas collection of infant feces: the first sample after birth and once a week during the period of hospitalization of the baby (i.e. 5 to 8 samples per infant) and a sample collected at the corrected age of 1 year and 2 years (i.e. 8 to 10 samples per infant). Associations between clinical metadata, dietary profiles and milk composition, and microbial community abundance will be investigate by Multivariate Association with Linear Models (MaAslin) and by applying Markov Decision Process (MDPs) to take into account the analysis of microbiota dynamics
Dietary profile and gut microbia composition | at 1 year of corrected age
  Correlation between 1-y infant dietary profile and 1-y infant gut microbiota composition. Associations between infant dietary profiles and microbial community abundance will be investigate by Multivariate Association with Linear Models (MaAslin) and by applying Markov Decision Process (MDPs) to take into account the analysis of microbiota dynamics
Dietary profile and gut microbia composition | at 2 years of corrected age
  Correlation between 1-y infant dietary profile and 2-y infant gut microbiota composition. Associations between infant dietary profiles and microbial community abundance will be investigate by Multivariate Association with Linear Models (MaAslin) and by applying Markov Decision Process (MDPs) to take into account the analysis of microbiota dynamics
Gut microbia | at 1 year of corrected age
  Functional activity of gut microbiota (in vitro test using 1-y infant fecal samples). Endocrine and barrier function responses of an in vitro tricellular model of intestinal epithelium (including enterocytes, mucin-secreting cells and entero-endocrine cells) to the stimulation by fecal water from 1-y infant feces will be characterized.
Gut microbia | at 2 years of corrected age
  Functional activity of gut microbiota (in vitro test using 1-y infant fecal samples). Endocrine and barrier function responses of an in vitro tricellular model of intestinal epithelium (including enterocytes, mucin-secreting cells and entero-endocrine cells) to the stimulation by fecal water from 1-y infant feces will be characterized.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes - Hôpital Sud, Rennes, France